CLINICAL TRIAL: NCT06996301
Title: Clinical Validity and Utility of PCR Compared to Conventional Culture and Sensitivity Testing for the Management of Complicated Urinary Tract Infections in Adults.
Brief Title: Clinical Utility of a PCR Compared to Culture and Sensitivity Testing for the Management of cUTI in Adults.
Acronym: PCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Doc Lab Inc (Industry)
Collaborators: Dicentra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 22-UPHUV-01
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-07

CONDITIONS: Urinary Tract Infection Complicated; Urinary Tract Infection (cUTI); Urinary Tract Infection (Diagnosis)
Keywords: Complicated urinary tract infection (cUTI); Polymerase Chain Reaction (PCR) diagnostic; Urine culture and sensitivity (C&S) testing; Favorable Clinical Outcomes (FCl); Turnaround Time; Randomized Controlled Trial (RCT); Treatment Outcome
MeSH Terms: conditions — Urinary Tract Infections; Disease; Pathologic Complete Response; Hypersensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- PCR Arm (Other): Treatment guided by the PCR results
  Interventions: Diagnostic Test: Treatment guided by the PCR results
- C&S Arm (Other): Treatment guided by the C&S results
  Interventions: Diagnostic Test: Treatment guided by the C&S results

INTERVENTIONS:
Diagnostic Test: Treatment guided by the PCR results — Patients receive treatment prescribed by a blinded clinician, based solely on the PCR diagnostic results
  Arms: PCR Arm
Diagnostic Test: Treatment guided by the C&S results — Patients receive treatment prescribed by a blinded investigator (clinician), based solely on the C&S diagnostic results.
  Arms: C&S Arm

SUMMARY:
Complicated urinary tract infections (cUTIs) often lead to the overuse of empiric antibiotics, risking inappropriate treatment and contributing to antimicrobial resistance. This randomized, multi-center, investigator-blinded clinical trial is the first global head-to-head comparison of molecular diagnostic testing (Polymerase Chain Reaction : PCR) versus conventional culture and sensitivity (C&S) for managing cUTIs in adults.

Conducted across six U.S. clinical sites, the study aimed to evaluate the clinical utility of PCR-guided treatment relative to C&S-guided care. Eligible adult patients were randomized 1:1 into two diagnostic arms-PCR or C&S-after providing informed consent. Urine samples were collected before randomization, tested by both methods, but clinicians remained blinded to the comparator results to avoid bias. Treatment decisions were based only on the assigned test results.

Urine was collected at baseline (Day 1) and at end-of-study (Day 28). Samples were processed centrally: the PCR method (DocLab UTM 2.0) detected 28 uropathogens and 16 antibiotic resistance gene classes; C&S testing quantified bacterial loads and assessed antimicrobial susceptibility using standard thresholds (≥10⁵ CFU/mL).

The primary endpoint was the number of patients in each arm achieving a Favorable Clinical Outcome (FCl) at Day 28, defined as either:

* Clinical Cure (complete symptom resolution requiring no further antibiotics), or
* Clinical Improvement (partial symptom resolution without new symptoms or IV antibiotics).

Secondary endpoints included:

* Microbiological eradication at EOS (via C&S and PCR).
* Clinician satisfaction with diagnostic usefulness and result clarity.
* Turnaround time comparison between PCR and C&S.
* Concordance analysis of test results between PCR and C&S.
* FCl rates in discordant cases, where PCR and C&S results disagreed.

DETAILED DESCRIPTION:
Study Overview:

Complicated urinary tract infections (cUTIs) remain a significant clinical challenge, often prompting empiric antibiotic use that may result in inappropriate therapy, antimicrobial overuse, and treatment failure. This study aimed to evaluate the clinical utility of molecular diagnostics (PCR) versus Conventional culture and sensitivity (C&S) methods in managing cUTIs, with the goal of identifying more effective patient management strategies.

This was a randomized, parallel-group, investigator-blinded, multi-center clinical trial conducted across six sites in the United States. Adults meeting all inclusion and no exclusion criteria who provided informed consent were randomized 1:1 into two arms: PCR-guided therapy and C&S-guided therapy. Each participant provided a urine sample before randomization, which was tested using both PCR and C&S. However, treating investigators remained blinded to the comparator test results throughout the study to ensure unbiased clinical decision-making.

Study Protocol:

Urine specimens were collected using a clean-catch midstream method at two time points: Day 1 (baseline) and Day 28 (end of study, EOS). Samples were refrigerated at 2-8°C and processed at a central lab. All specimens were split for parallel testing using:

* PCR (DocLab UTM 2.0): A qualitative panel targeting 28 uropathogen species and 16 antimicrobial resistance gene classes via QuantStudio 7/12 and KingFisher platforms.
* Conventional C&S: Quantitative bacterial culture and sensitivity testing to identify uropathogens and assess resistance profiles, with a detection threshold of ≥10⁵ CFU/mL.

Blinding and Treatment Allocation:

Participants were treated based exclusively on the test result assigned by randomization (PCR or C&S). Comparator test results were withheld from clinicians until after the study concluded.

The primary endpoint was the number (and percentage) of subjects in each study arm with favorable clinical outcomes (FCl) at the EOS visit. The FCl was defined as a patient's clinical response, assessed by the treating investigator, indicating either clinical improvement or cure. Clinical improvement was defined as the resolution of at least one symptom of cUTI present at baseline, absence of new cUTI symptoms, and/or avoidance of parenteral antibiotic therapy following randomization. Clinical cure was defined as the complete resolution of all acute signs and symptoms of cUTI present at baseline, to the extent that no further antimicrobial therapy (either IV or oral) was required for the treatment of the cUTI.

The secondary endpoint included several assessments:

* Number (and percentage) of subjects with microbiological eradication at the EOS, defined as achieving a quantitative urine culture at the EOS indicating a reduction of all uro-pathogens present at baseline to <10^5 colony forming unit per milliliter (CFU/mL) and the absence of baseline pathogens detected by EOS urine PCR (Cq > 33);
* Subjective measurement of treating investigator satisfaction score through a questionnaire (5 questions) at EOS, evaluated factors such as (1) result availability/timeliness, (2) clarity of result interpretation, (3) clinical decision-making utility, (4) overall test satisfaction, and (5) perceived impact on patient outcomes versus comparator.
* Comparison of turnaround time between molecular diagnostic procedures and conventional diagnostic
* Overall agreeability between the diagnostic results generated by PCR versus C&S as assessed by discordant analysis
* Assessment of the favorable clinical outcome of patients with discordant results [PCR(+), CS(-) and PCR(-), CS(+)]

ELIGIBILITY:
Inclusion Criteria:

* I1. At least 18 years of age at the time of consent
* I2. Presenting at least two of the following new, persistent or worsening cUTI signs and symptoms at screening visit: a) fever (temperature >38 degrees Celsius or >100.4 degrees Fahrenheit), hypothermia (temperature <35.5 degrees Celsius or <95.9 degrees Fahrenheit), rigors, or chills b) dysuria, urinary frequency, urgency, or hematuria c) suprapubic pain or pelvic pain d) costovertebral angle (CVA) tenderness e) nausea or vomiting f) radiographic evidence of pyelonephritis g) leukocytosis
* I3. Urine specimen with evidence of pyuria a) dipstick analysis positive for nitrite and/or leukocyte esterase, or; b) ≥10 white blood cells (WBCs) per cubic millimeter [mm3], or; c) ≥10 WBCs per high power field (hpf), or; d) clinically suspected pyuria (e.g. change in urine color, sediment in urine, or foul-smelling urine)
* I4. Having cUTI that requires microbiological diagnosis and treatment as suspected by the Investigator
* I5. Presenting active UTI that failed to resolve on first-line therapy or identified as a high-risk* patient population; *High-risk patient population include those who are elderly (≥65years), male, pregnant, having recurrent UTI (≥3/year), with underlying co-morbidities (e.g. diabetes, immunosuppression, or CKD), or with known functional and anatomical abnormalities of the urinary tract (e.g. stones, stents, recent instrumentation, indwelling catheters, neurogenic bladder, or PKD)
* I6. Able to provide at least 8 mL urine at visit 1 and 3
* I7. Willing to abstain from sexual intercourse or use condoms during any sexual contact until the End-of-Study (EOS) visit is complete
* I8. Willing to comply with protocol requirements, including availability for follow-up for the duration of the study

Exclusion Criteria:

* E1. Unable or unwilling to provide written informed consent
* E2. Unable to read and write in English (surveys are not available or validated in any other language than English)
* E3. Currently participating in or has participated in an interventional clinical trial with an investigational product or device within 30 days prior to the Screening Visit
* E4. Currently on or chronic use of any antibiotics for any clinical indication, other than UTI
* E5. Receipt of any dose of a potentially therapeutic oral or systemic antibiotics for the treatment of UTI within 48 hours before the study baseline urine is obtained
* E6.Pregnant women with known fetal congenital anomaly (e.g., genetic abnormality or major congenital malformation) based on antenatal ultrasound
* E7. Any rapidly progressing disease or immediately life-threatening illness, including acute hepatic failure, or respiratory failure
* E8. Medical condition or other factor that in the judgment of the investigator might affect ability to comply with procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roel Chavez, Study Chair — Doc Lab Inc; Thomas K Huard, PhD, Principal Investigator — MED-US Consulting, LLC
Locations (6):
- United States (6):
  - Silicon Valley Medical Development, San Jose, California
  - Albany Urology Clinic & Surgery Center, Albany, Georgia
  - Augusta Urology Associates, Evans, Georgia
  - Colquitt Regional Medical Center, Moultrie, Georgia
  - Phoenix Urology of St Joseph, Saint Joseph, Missouri
  - Norman Urology Associates, Norman, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between July 2023 and April 2024, 824 patients were screened, and 773 were randomized with informed consent. Both PCR and C&S testing were performed for all enrolled participants (n = 773) before randomization into one of the two study arms
Period: Overall Study
Arm/Group | PCR Arm | C&S Arm
Started | 397 | 376
Completed | 193 | 169
Not Completed | 204 | 207
Not completed — Patients with negative microbiological evidence by both diagnostic methods | 54 | 54
Not completed — Patients with discordant diagnostic results | 107 | 90
Not completed — Lost to Follow-up | 31 | 56
Not completed — Withdrawal by Subject | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCR Arm | C&S Arm | Total
Number analyzed (Participants) | 397 | 376 | 773
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 49 | 101
  >=65 years | 345 | 327 | 672
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 263 | 535
  Male | 125 | 113 | 238
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Favorable Clinical Outcomes (FCl)
Description: The number (and percentage) of subjects in each study arm with favorable clinical outcomes (FCl) at the EOS visit. The FCl was defined as a patient's clinical response, assessed by the treating investigator, indicating either clinical improvement or cure. Clinical improvement was defined as the resolution of at least one symptom of cUTI present at baseline, absence of new cUTI symptoms, and/or avoidance of parenteral antibiotic therapy following randomization. Clinical cure was defined as the complete resolution of all acute signs and symptoms of cUTI present at baseline, to the extent that no further antimicrobial therapy (either IV or oral) was required for the treatment of the cUTI.
Time Frame: at End Of Study (EOS) visit (Day 28)
Population: EOS Population: This group included all enrolled patients who completed the study procedures, including the treating investigators' evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | PCR Arm | C&S Arm
Number analyzed (Participants) | 193 | 169
Participants | 170 | 132

2. Secondary Outcome: Microbiological Eradication
Description: Number (and percentage) of subjects with microbiological eradication at the EOS, defined as achieving a quantitative urine culture at the EOS indicating a reduction of all uro-pathogens present at baseline to <10^5 colony forming unit per milliliter (CFU/mL) and the absence of baseline pathogens detected by EOS urine PCR (Cq > 33)
Time Frame: at End Of Study (EOS) visit (Day 28)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PCR Arm | C&S Arm
Number analyzed (Participants) | 193 | 169
Participants | 120 | 95

3. Secondary Outcome: Treating Investigator Satisfaction Score
Description: Subjective measurement of treating investigator satisfaction score through a questionnaire (5 questions) at EOS, evaluated factors such as (1) result availability/timeliness, (2) clarity of result interpretation, (3) clinical decision-making utility, (4) overall test satisfaction, and (5) perceived impact on patient outcomes versus comparator.
  Scale information Score Interpretation: Each item scored 1-5; higher scores reflect greater diagnostic and therapeutic value.
  Total score meaning:
  * ≥20: Good clinical utility.
  * 10-19: Moderate utility.
  * 1-9: Poor utility.
Time Frame: at End Of Study (EOS) visit (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale (1-25)
Arm/Group | PCR Arm | C&S Arm
Number analyzed (Participants) | 193 | 169
score on a scale (1-25) | 23.95 (1.96) | 20.64 (4.12)

4. Secondary Outcome: Turnaround Time
Description: Comparison of turnaround time between molecular diagnostic procedures and conventional diagnostic
Time Frame: at End Of Study (EOS) visit (Day 28)
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Arm/Group | PCR Arm | C&S Arm
Number analyzed (Participants) | 193 | 169
hours | 49.68 [2.41 to 152.53] | 104.4 [48.21 to 592.53]

5. Secondary Outcome: Overall Agreeability
Description: Overall agreeability between the diagnostic results generated by PCR versus C&S as assessed by discordant analysis
Time Frame: at End Of Study (EOS) visit (Day 28)
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | PCR Arm
Number analyzed (Participants) | 193
percentage
  Sensitivity % | 88.6
  Specificity % | 62.91

6. Secondary Outcome: Favorable Clinical Outcome of Patients With Discordant Results
Description: Assessment of the favorable clinical outcome of patients with discordant results [PCR(+), CS(-) and PCR(-), CS(+)] Patients with discordant results [PCR(+), CS(-) and PCR(-), CS(+)] were excluded from the primary endpoint analysis and their outcome is presented here as a secondary analysis
Time Frame: at End Of Study (EOS) visit (Day 28)
Population: Patients with discordant results PCR Arm : PCR(+), CS(-) & C&S Arm : PCR(-), CS(+)
  Note:
  PCR Arm: No patients were identified as PCR(-), CS(+). C&S Arm: A total of 68 patients were PCR(+), CS(-). Their clinical outcomes were not reported in this study, as they were managed with empiric therapy rather than pathogen-directed treatment.
Measure: Count of Participants; unit: Participants
Groups:
- PCR Arm : PCR(+), CS(-): Treatment guided by the PCR results
- C&S Arm : PCR(-), CS(+): Treatment guided by the C&S results
Arm/Group | PCR Arm : PCR(+), CS(-) | C&S Arm : PCR(-), CS(+)
Number analyzed (Participants) | 102 | 14
Participants | 79 | 10

ADVERSE EVENTS:
Time Frame: Day 1 (baseline) and Day 28 (end of study, EOS)
Description: All events will be managed promptly and reported in compliance with all applicable regulations and guidelines.
Arm/Group | PCR Arm | C&S Arm
All-Cause Mortality (participants affected / at risk) | 0/236 | 0/232
Serious Adverse Events (participants affected / at risk) | 0/236 | 0/232
Other Adverse Events (participants affected / at risk) | 0/236 | 0/232

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT06996301/Prot_SAP_ICF_001.pdf